CLINICAL TRIAL: NCT06025253
Title: Prophylactic Single-Use Negative Pressure Wound Therapy Devices for Closed Incision Major Amputations
Brief Title: PINTA - Prophylactic Incisional Negative Pressure Therapy for Major Amputations
Acronym: PINTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCSI- PINTA
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-03

CONDITIONS: Wound Surgical; Wound Infection; Cosmesis
Keywords: Negative Pressure Wound Therapy; Surgical Site Infection; Post-operative Complications; Health Economics; CoPaQ; WoundQol
MeSH Terms: conditions — Surgical Wound; Wound Infection; Surgical Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative Pressure Wound Therapy. (Experimental): Application of a negative wound pressure therapy dressing to the wound post major lower extremity amputation
  Interventions: Device: Negative Pressure Wound Therapy
- Standard Wound dressing (Active Comparator): Application of sterile standard gauze dressing to the wound post major lower extremity amputation
  Interventions: Device: Standard Wound Dressing

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — Application of negative-pressure wound therapy (NPWT) post major lower extremity amputation
  Arms: Negative Pressure Wound Therapy.
Device: Standard Wound Dressing — Application of standard wound dressing post major lower extremity amputation
  Arms: Standard Wound dressing

SUMMARY:
Post-operative wound issues in abdominal surgery have a significant impact on patient outcomes. This study is taking place to investigate if Negative Pressure Wound Therapy (NPWT) dressings reduces Surgical Site Infections, post surgical complications and improves scar appearance compared to standard dressings.

DETAILED DESCRIPTION:
Many factors influence the risk of wound complications. Notably, the presence of unreconstructed proximal occlusive arterial disease is a major influence on stump healing. Patient factors such as smoking, diabetes, obesity, malnutrition and chronic kidney disease are non-modifiable, particularly in the short-term setting. However, surgical factors may be altered in an effort to reduce the risk of wound complications.

One option amenable to alteration is what dressing is applied to the closed incision upon procedure completion. The type of dressing may influence factors such as bacterial access to the wound, the development of collections of blood or fluid in the wound or fluid oozing from the wound. Collectively, these wound factors increase the risk of wound infection. Therefore, dressings which reduce these factors have the potential to reduce wound breakdown, thereby reducing the burden for patients and healthcare systems.

The investigators propose to conduct a multicentre randomised controlled trial comparing prophylactic single-use negative pressure wound therapy with standard dressings in patients with a closed incision following major lower extremity amputation in terms of SSI incidence, wound healing complications and scar appearance, patient quality of life and financial impact on the patient and healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older;
* Patients undergoing major lower extremity amputation, including below-knee amputation, through-knee amputation and above-knee amputation, for any indication;
* Patients with primary closure of the surgical incision using either interrupted or continuous sutures

Exclusion Criteria:

* Patients <18 years;
* Women who are pregnant and/or breast-feeding;
* Patients with amputations performed without primary skin closure, including guillotine amputations, amputations deliberately left open for drainage purposes and amputations with soft tissues defects at the stump;
* Patients with amputations where skin glue is the only means of skin closure
* Patients with a clinically absent femoral pulse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 728 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Presence of wound complications following amputation between NPWT and standard dressings | 1 month following surgery
  Infection(deep or superficial), wound dehiscence, partial (fascia intact), complete (fascia breached), seroma, haematoma or stump necrosis.

SECONDARY OUTCOMES:
Number of days to discharge | 6 months following surgery
  Length of time patient is in hospital from date of surgery to date of discharge
Rate of re-admission | 1 Month following surgery
  Number of re-admissions to the hospital from date of surgery
Health-related quality of life with the EuroQol-5 dimensions five level index questionnaire (EQ-5D-5L) | Baseline
  The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)
Health-related quality of life with the EuroQol-5 dimensions five level index questionnaire (EQ-5D-5L) | 1 month following surgery
  The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)
Health-related quality of life with the EuroQol-5 dimensions five level index questionnaire (EQ-5D-5L) | 3 months following surgery
  The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)
Health-related quality of life with the EuroQol-5 dimensions five level index questionnaire (EQ-5D-5L) | 6 months following surgery
  The questionnaire covers five dimensions of health: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The raw scores are also converted to an EQ-5D index value using a scoring algorithm (British tariff) ranging from -0.594 (worst perceived health state) to 1.00 (best perceived health state)
Wound-QoL (Questionnaire on quality of life with chronic wounds) | 1 month following surgery
  Wound-QoL (Questionnaire on quality of life with chronic wounds) measures the disease-specific, health-related quality of life of patients with chronic wounds. It can be used in clinical and observational studies as well as in daily practice. The primary endpoint is the reduction of more than 0.4 points in the overall score of the Wound-Qol quality of life questionnaire between D0 and D14.
Wound-QoL (Questionnaire on quality of life with chronic wounds) | 3 months following surgery
  Wound-QoL (Questionnaire on quality of life with chronic wounds) measures the disease-specific, health-related quality of life of patients with chronic wounds. It can be used in clinical and observational studies as well as in daily practice. The primary endpoint is the reduction of more than 0.4 points in the overall score of the Wound-Qol quality of life questionnaire between D0 and D14.
Wound-QoL (Questionnaire on quality of life with chronic wounds) | 6 months following surgery
  Wound-QoL (Questionnaire on quality of life with chronic wounds) measures the disease-specific, health-related quality of life of patients with chronic wounds. It can be used in clinical and observational studies as well as in daily practice. The primary endpoint is the reduction of more than 0.4 points in the overall score of the Wound-Qol quality of life questionnaire between D0 and D14.
Health-related out-of- Pocket Costs assessed using the Costs for Patients Questionnaire (CoPaQ) | 1 Month following surgery
  The CoPaQ measures patient and caregivers out-of-pocket expenses (direct and indirect) associated with a health condition
Health-related out-of- Pocket Costs assessed using the Costs for Patients Questionnaire (CoPaQ) | 3 Months following surgery
  The CoPaQ measures patient and caregivers out-of-pocket expenses (direct and indirect) associated with a health condition
Health-related out-of- Pocket Costs assessed using the Costs for Patients Questionnaire (CoPaQ) | 6 Months following surgery
  The CoPaQ measures patient and caregivers out-of-pocket expenses (direct and indirect) associated with a health condition
Rate of Re-operation | 1 Month following surgery
  Number of re-operations undertaken from date of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Walsh, Prof, Principal Investigator — University Hospital Galway (UHG)
Locations (7):
- Ireland (7):
  - Beaumont Hospital, Beaumont rd,Dublin 9, D09V2N0, Dublin
  - St Jamess Hospital, Dublin
  - St Vincents University Hospital, Dublin
  - Tallaght University Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Limerick, Limerick
  - University Hospital Waterford, Waterford

IPD SHARING:
Plan to Share IPD: No